CLINICAL TRIAL: NCT02824055
Title: A Study to Evaluate The Effects of RO5545965 in Participants With Negative Symptoms of Schizophrenia Treated With Antipsychotics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BP29904
Record Dates: First submitted 2016-06-21; First posted 2016-07-06 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Placebo first; then RO5545965 15 mg; then RO5545965 5mg (Placebo Comparator): Participants will receive placebo matched to RO5545965 capsules orally daily from Weeks 1 to 3 in first intervention period; then RO5545965 15 mg capsules (5 mg for 3 days, 10 mg for 3 days and 15 mg for 15 days) orally daily from Weeks 6 to 8 in second intervention period; followed by RO5545965 5 mg capsules orally daily from Weeks 11 to 13 in third intervention period. A washout period of minimum 14 days will be maintained between each period.
  Interventions: Drug: Placebo; Drug: RO5545965
- Placebo first; then RO5545965 5 mg; then RO5545965 15 mg (Placebo Comparator): Participants will receive placebo matched to RO5545965 capsules orally daily from Weeks 1 to 3 in first intervention period; then RO5545965 5 mg capsules orally daily from Weeks 6 to 8 in second intervention period; followed by RO5545965 15 mg capsules (5 mg for 3 days, 10 mg for 3 days and 15 mg for 15 days) orally daily from Weeks 11 to 13 in third intervention period. A washout period of minimum 14 days will be maintained between each period.
  Interventions: Drug: Placebo; Drug: RO5545965
- RO5545965 15 mg first; then Placebo; then RO5545965 5 mg (Experimental): Participants will receive RO5545965 15 mg capsules (5 mg for 3 days, 10 mg for 3 days and 15 mg for 15 days) orally daily from Weeks 1 to 3 in first intervention period; then placebo matched to RO5545965 capsules orally daily from Weeks 6 to 8 in second intervention period; followed by RO5545965 5 mg capsules orally daily from Weeks 11 to 13 in third intervention period. A washout period of minimum 14 days will be maintained between each period.
  Interventions: Drug: Placebo; Drug: RO5545965
- RO5545965 15 mg first; then RO5545965 5 mg; then Placebo (Experimental): Participants will receive RO5545965 15 mg capsules (5 mg for 3 days, 10 mg for 3 days and 15 mg for 15 days) orally daily from Weeks 1 to 3 in first intervention period; then RO5545965 5 mg capsules orally daily from Weeks 6 to 8 in second intervention period; followed by placebo matched to RO5545965 capsules orally daily from Weeks 11 to 13 in third intervention period. A washout period of minimum 14 days will be maintained between each period.
  Interventions: Drug: Placebo; Drug: RO5545965
- RO5545965 5 mg first; then Placebo; then RO5545965 15 mg (Experimental): Participants will receive RO5545965 5 mg capsules orally daily from Weeks 1 to 3 in first intervention period; then placebo matched to RO5545965 capsules orally daily from Weeks 6 to 8 in second intervention period; followed by RO5545965 15 mg capsules (5 mg for 3 days, 10 mg for 3 days and 15 mg for 15 days) orally daily from Weeks 11 to 13 in third intervention period. A washout period of minimum 14 days will be maintained between each period.
  Interventions: Drug: Placebo; Drug: RO5545965
- RO5545965 5 mg first; then RO5545965 15 mg; then Placebo (Experimental): Participants will receive RO5545965 5 mg capsules orally daily from Weeks 1 to 3 in first intervention period; then RO5545965 15 mg capsules (5 mg for 3 days, 10 mg for 3 days and 15 mg for 15 days) orally daily from Weeks 6 to 8 in second intervention period; followed by placebo matched to RO5545965 capsules orally daily from Weeks 11 to 13 in third intervention period. A washout period of minimum 14 days will be maintained between each period.
  Interventions: Drug: Placebo; Drug: RO5545965

INTERVENTIONS:
Drug: Placebo — Participants will receive placebo matched to RO5545965 capsules orally daily in any of the three intervention period.
Drug: RO5545965 — Participants will receive RO5545965 5 mg capsules or RO5545965 15 mg capsules (5 mg for 3 days, 10 mg for 3 days and 15 mg for 15 days) orally daily in any of the three intervention period.

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, three period crossover study to evaluate the effects of RO5545965 on the functioning of key brain circuitry involved in negative symptoms using functional magnetic resonance imaging (fMRI) and reward-based learning in stable participants with mild to moderate negative symptoms of schizophrenia treated with antipsychotics. Participants will be randomized to one of six different sequences during which each participant will receive three 3-week treatment courses with RO5545965 5 milligrams (mg), RO5545965 15 mg and placebo. Each treatment period will be separated by a washout period of 14 days. Total duration of study will be approximately 17 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A diagnostic and statistical manual of mental disorders-5 (DSM-5) diagnosis of schizophrenia as established by structured clinical interview for DSM-5-clinical trial (SCID-5-CT) at screening
* Participants with no hospitalization for worsening of schizophrenia within 3 months prior to screening
* Male and female participants with no childbearing capacity; females must be either surgically sterile or postmenopausal for at least 1 year
* Body mass index (BMI) greater than (>) 18.5 kilograms per square meter (kg/m^2) and less than (<) 35 kg/m^2
* Fluent in English, even if English is not the primary language
* Participants with clinical global impression-severity (CGI-S) score greater than or equal to (>/=) 3 (mildly ill)
* Participants with a score of less than or equal to (</=) 4 (moderate) on positive and negative syndrome scale (PANSS) items P7 (hostility), G8 (uncooperativeness) and G6 (depression)
* Participants with PANSS negative symptom factor score >/=18
* Participants with calgary depression rating scale for schizophrenia (CDSS) score </=8
* Participants on stable treatment, that is 6 weeks without change, with no more than two antipsychotics prior to screening

Exclusion Criteria:

* Moderate to severe substance use disorder within 6 months as defined by DSM-5
* Positive urine drug screen for amphetamines, methamphetamines, opiates, buprenorphine, methadone, cannabinoids, cocaine and barbiturates
* Participants at significant risk of suicide or harming him or herself or others according to the Investigator's judgment
* History of neuroleptic malignant syndrome
* A prior or current general medical condition that might be impairing cognition or other psychiatric functioning
* A movement disorder due to antipsychotic treatment not currently controlled with anti-extrapyramidal symptoms (anti-EPS) treatment or another movement disorder which might affect the ratings on the EPS scales
* Participants with a score >2 (mild) in any of the four CGI-S items of the extrapyramidal symptom rating scale (ESRS-A)
* History of human immunodeficiency virus (HIV) infection, Hepatitis B, or Hepatitis C infection
* QTcF interval >450 milliseconds (msec) (470 msec for females) or other significant abnormality on screening electrocardiogram (ECG) based on centralized reading
* Clinically significant abnormalities in laboratory safety test results
* Significant or unstable physical condition
* Receipt of an investigational drug within 90 days or 5 times the half-life of the investigational drug, whatever is longer, prior to screening
* Previously received RO5545965
* Electroconvulsive treatment (ECT) within 6 months prior to screening
* Current or 6 months prior to screening treatment with olanzapine or clozapine
* Change in benzodiazepine or sleep medication regimen within 2 weeks prior to screening
* Change in anti-EPS medication within two weeks prior to screening
* Use of prohibited medications taken within 14 days or within 5 times the elimination half-life of the medication before the first study drug administration
* Use of any strong or moderate inhibitor of cytochrome P 450 3A (CYP3A) or CYP2C8 and any inducer of CYP3A within 14 days or within 5 times the elimination half-life of the medication (whichever is longer) before the first study drug administration
* Use of any other nutrients known to modulate CYP3A activity within 1 week before the first study drug administration

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
Apparent volume of distribution (Vz/F) | Pre-dose on Days 8, 15, 22, 43, 50, 57, 78, 85 and 96; additional 2 hour post-dose on Days 15, 50, and 85
Activity of the ventral striatum during reward expectation in a monetary incentive delay fMRI task as measured by blood oxygen level dependent (BOLD) activity | Baseline (Day 1) up to end of study (up to 17 weeks)
Performance in reward based learning tasks as measured by the working memory reinforcement learning task | Day 22 up to Day 92
Performance in reward based learning tasks as measured by the effort cost/benefit tradeoff task | Day 22 up to Day 92
Apparent oral clearance (CL/F) | Pre-dose on Days 8, 15, 22, 43, 50, 57, 78, 85 and 96; additional 2 hour post-dose on Days 15, 50, and 85

SECONDARY OUTCOMES:
Activity in the dorsolateral prefrontal cortex in the N-back working memory task as measured by BOLD activity | Baseline (Day 1) up to end of study (up to 17 weeks)
Cerebral blood flow in key brain areas (ventral striatum, orbitofrontal cortex) implicated in the etiology of negative symptoms as measured by arterial spin labeling (ASL) | Baseline (Day 1) up to end of study (up to 17 weeks)
Overall symptoms score of schizophrenia based on total PANSS | Baseline (Day 1), Days 22, 57, and 92
Symptom domains of schizophrenia based on PANSS factor subscales | Baseline (Day 1), Days 22, 57, and 92
Negative symptoms score of schizophrenia based on brief negative symptom scale (BNSS) | Baseline (Day 1), Days 22, 57, and 92
Overall clinical status based on CGI-S scores | Baseline (Day 1), Days 22, 57, and 92
Overall clinical status based on CGI-Improvement (CGI-I) score | Baseline (Day 1), Days 22, 57, and 92
Overall global impression of negative symptoms based on CGI-S negative symptoms | Baseline (Day 1), Days 22, 57, and 92
Overall global impression of negative symptoms based on CGI-I negative symptoms | Baseline (Day 1), Days 22, 57, and 92
Area under the concentration-time curve (AUC) | Pre-dose on Days 8, 15, 22, 43, 50, 57, 78, 85 and 96; additional 2 hour post-dose on Days 15, 50, and 85
Maximum observed plasma concentration (Cmax) | Pre-dose on Days 8, 15, 22, 43, 50, 57, 78, 85 and 96; additional 2 hour post-dose on Days 15, 50, and 85
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Screening (Day -15 to Day -1) up to end of study (up to 17 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (3):
  - CNS Network, Garden Grove, California
  - Parexel California Clinical Trials Medical Group, Glendale, California
  - St Louis Clinical Trials, St Louis, Missouri

REFERENCES:
- [Derived] Omlor W, Cecere G, Huang GY, Spiller T, Misra AR, Rabe F, Kallen N, Kirschner M, Surbeck W, Burrer A, Garibaldi G, Holiga S, Dukart J, Umbricht D, Homan P. Exploratory analysis of the relationship between striatal connectivity and apathy during phosphodiesterase 10 inhibition in schizophrenia: findings from a randomized crossover trial. BMC Med. 2025 Mar 28;23(1):187. doi: 10.1186/s12916-025-04004-2. PMID 40155941
- [Derived] Umbricht D, Cheng WY, Lipsmeier F, Bamdadian A, Lindemann M. Deep Learning-Based Human Activity Recognition for Continuous Activity and Gesture Monitoring for Schizophrenia Patients With Negative Symptoms. Front Psychiatry. 2020 Sep 16;11:574375. doi: 10.3389/fpsyt.2020.574375. eCollection 2020. PMID 33192706